CLINICAL TRIAL: NCT01466218
Title: Pulmonary Abnormalities, Diastolic Dysfunction, and World Trade Center Exposure: Implications for Diagnosis and Treatment
Brief Title: World Trade Center (WTC) CHEST
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: GCO 11-0618; BAA (2011-Q-13340) (Other: NIOSH)
Record Dates: First submitted 2011-10-28; First posted 2011-11-07 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease; Cardiac Disease; Cardiopulmonary Disease; Obstructive Sleep Apnea; Cardiovascular Disease
Keywords: pulmonary function abnormalities; pulmonary disease; cardiac disease; cardiopulmonary disease; obstructive sleep apnea; OSA; cardiovascular disease; CVD; particulate matter
MeSH Terms: conditions — Lung Diseases; Heart Diseases; Pulmonary Heart Disease; Sleep Apnea, Obstructive; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- WTC Volunteers and Workers: Any current participant of the World Trade Center Health Program-Clinical Center of Excellence, formerly known as World Trade Center Medical Monitoring and Treatment Program

SUMMARY:
This project will evaluate the effects of World Trade Center (WTC) exposure in WTC responders 10-13 years following the events of 9/11. Prior studies have described persistent pulmonary function abnormalities in a significant portion of responders. The investigators study seeks to examine the relationship between pulmonary function abnormalities and other markers of chronic cardiopulmonary disease and further elucidate the pathophysiologic effects of exposure to inhaled particulate matter (PM) on 9/11. This study will provide critical information regarding risk of exposure to PM, risk factors for disease and potential for improvements in diagnosis and treatment.

DETAILED DESCRIPTION:
Serious illness and injury following the September 11, 2001 (9/11) attacks on the World Trade Center (WTC) affects thousands of responders who worked on the WTC rescue and recovery effort. During this time, these individuals sustained exposure to a vast array of environmental toxins and physical hazards. The population of survivors presents a unique opportunity to rigorously examine the effects of inhaled particulate matter on risk of persistent pulmonary and chronic cardiopulmonary disease.

Original reports of 9,500 WTC responders examined between July 2002 and April 2004, noted abnormal pulmonary function results in one-third of participants. Further studies of this population have demonstrated persistent changes in pulmonary function tests 9 years after exposure (2010 Annual Report on 9/11 Health). Numerous complex interactions between pulmonary and cardiovascular systems exist. In fact, at the molecular level, evidence supports an integral role for reactive oxygen species (ROS)-dependent pathways in the instigation of pulmonary oxidative stress, systemic pro-inflammatory responses, vascular dysfunction and atherosclerosis.

Studies in animals have shown that inhalation of particles can lead to weakening of the heart muscle. In addition, patients who have developed pulmonary disease from inhalation of particulate matter may develop increased pressures in the pulmonary arteries, as well as dysfunction of the right ventricle of the heart. Finally, patients who have suffered blockage of the coronary arteries may exhibit abnormalities in the heart function that may be detected by an echocardiogram.

Preliminary work by our group revealed echocardiographic evidence of cardiac abnormalities in a subset of 1190 WTC responders. Diastolic dysfunction, or impaired ventricular relaxation, is known to accompany aging and is associated with hypertensive heart disease. In our analysis of subjects < 50 years of age, BMI < 30, and lacking a diagnosis of hypertension, the investigators found a prevalence of diastolic dysfunction of 47%. Importantly, when the population was narrowed to exclude former or current smokers, and those with LV abnormalities, 12% had abnormalities of RV diastolic function. The investigators propose to analyze the relationship between pulmonary function abnormalities and evidence of diastolic dysfunction.

Persuasive data implicates obstructive sleep apnea (OSA) in the development of hypertension, arrhythmias, vascular dysfunction and cardiac disease. Webber et al demonstrated an increased prevalence of obstructive sleep apnea (OSA) among firefighters exposed to the WTC disaster, and our group has demonstrated a similar prevalence of screen positive for OSA among 2500 law enforcement officers present at Ground Zero. The relationship between OSA and risk of cardiac disease involves similar pathophysiologic pathways including inflammation and impaired vascular reactivity.

In addition to the traditional risk factors for cardiovascular disease (CVD), studies have indicated that exposure to inhalation of particulate matter (PM) contribute to CV morbidity and mortality. The 2010 American Heart Association Scientific Statement on Particulate Matter Air Pollution and Cardiovascular Disease provided compelling evidence of increased risk due to air pollution. Although the exact mechanisms by which PM cause these toxic effects are not adequately understood, and it is likely that different mechanisms are responsible for acute and chronic effects. In addition, PM consists of many different components, and different components may affect CVD by different mechanisms, such as electrophysiologic changes, inflammation, coagulation, endothelial cell function effects and atherosclerosis. In summary, thousands of WTC responders sustained exposure to thousands of tons of coarse and fine PM, cement dust, glass fibers, asbestos, lead, hydrochloric acid, polychlorinated biphenyls, organochlorine pesticides, and polychlorinated dioxins and furans. It is unknown to what extent the exposure to PM modified risk of developing atherosclerotic disease, in addition to the pulmonary effects and effects on cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* World Trade Center responders who are currently enrolled in the World Trade Center Health Program-Clinical Center of Excellence, formerly known as the WTC Medical Monitoring and Treatment Program
* Over the age of 39 years

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: World Trade Center rescue and recovery workers and volunteers who are enrolled in the World Trade Center Health Program-Clinical Center of Excellence, formerly known as the Medical Monitoring Treatment Program
Sampling Method: Non-Probability Sample
Enrollment: 1012 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Spirometry | day 1
  To evaluate the persistent longitudinal effects of pulmonary function abnormalities (spirometry) and additionally demonstrate prevalence of impaired DLCO in WTC responders.

SECONDARY OUTCOMES:
RV diastolic dysfunction | day 1
  To determine the relationship between pulmonary function abnormalities (spirometry and DLCO) and cardiac dysfunction using echocardiograms to measure right ventricular (RV) diastolic dysfunction.
LV diastolic function | day 1
  To evaluate the association between levels of exposure to inhaled particulate matter on cardiac dysfunction as measured by left ventricular (LV) diastolic function or evidence of subclinical atherosclerosis with high risk coronary calcium scores in WTC responders.
obstructive sleep apnea risk | day 1
  To determine the risks of developing obstructive sleep apnea (OSA) in the WTC responder population, and to evaluate the effect of OSA on mediating diastolic dysfunction.
microvascular and cardiovascular disease | day 1
  To demonstrate specific mediators and pathways that link effects of inhaled particulate matter to microvascular and cardiovascular disease. This objective will be explored using measurements of vascular reactivity (peripheral arterial tonometry) and serum inflammatory and hemostatic markers from blood stored at the initial monitoring visit, as well as current blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann McLaughlin, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Herbert R, Moline J, Skloot G, Metzger K, Baron S, Luft B, Markowitz S, Udasin I, Harrison D, Stein D, Todd A, Enright P, Stellman JM, Landrigan PJ, Levin SM. The World Trade Center disaster and the health of workers: five-year assessment of a unique medical screening program. Environ Health Perspect. 2006 Dec;114(12):1853-8. doi: 10.1289/ehp.9592. PMID 17185275
- [Background] 2010 Annual Report on 9/11 Health. Available at: www.nyc.gov/9-11HealthInfo.
- [Background] Dominici F, Peng RD, Bell ML, Pham L, McDermott A, Zeger SL, Samet JM. Fine particulate air pollution and hospital admission for cardiovascular and respiratory diseases. JAMA. 2006 Mar 8;295(10):1127-34. doi: 10.1001/jama.295.10.1127. PMID 16522832
- [Background] Pope CA 3rd, Hansen ML, Long RW, Nielsen KR, Eatough NL, Wilson WE, Eatough DJ. Ambient particulate air pollution, heart rate variability, and blood markers of inflammation in a panel of elderly subjects. Environ Health Perspect. 2004 Mar;112(3):339-45. doi: 10.1289/ehp.6588. PMID 14998750
- [Background] Brook RD, Franklin B, Cascio W, Hong Y, Howard G, Lipsett M, Luepker R, Mittleman M, Samet J, Smith SC Jr, Tager I; Expert Panel on Population and Prevention Science of the American Heart Association. Air pollution and cardiovascular disease: a statement for healthcare professionals from the Expert Panel on Population and Prevention Science of the American Heart Association. Circulation. 2004 Jun 1;109(21):2655-71. doi: 10.1161/01.CIR.0000128587.30041.C8. PMID 15173049
- [Background] Hamade AK, Tankersley CG. Interstrain variation in cardiac and respiratory adaptation to repeated ozone and particulate matter exposures. Am J Physiol Regul Integr Comp Physiol. 2009 Apr;296(4):R1202-15. doi: 10.1152/ajpregu.90808.2008. Epub 2009 Jan 21. PMID 19158411
- [Background] Tankersley CG, Champion HC, Takimoto E, Gabrielson K, Bedja D, Misra V, El-Haddad H, Rabold R, Mitzner W. Exposure to inhaled particulate matter impairs cardiac function in senescent mice. Am J Physiol Regul Integr Comp Physiol. 2008 Jul;295(1):R252-63. doi: 10.1152/ajpregu.00697.2007. Epub 2008 Apr 30. PMID 18448608
- [Background] Croft L, McLaughlin MA, Bander J, et al. First Documentation of Cardiac Dysfunction Following Exposure to the World Trade Center Disaster. JACC. 2010;55:A86.E810.
- [Background] Shamsuzzaman AS, Gersh BJ, Somers VK. Obstructive sleep apnea: implications for cardiac and vascular disease. JAMA. 2003 Oct 8;290(14):1906-14. doi: 10.1001/jama.290.14.1906. PMID 14532320
- [Background] Webber MP, Lee R, Soo J, Gustave J, Hall CB, Kelly K, Prezant D. Prevalence and incidence of high risk for obstructive sleep apnea in World Trade Center-exposed rescue/recovery workers. Sleep Breath. 2011 Sep;15(3):283-94. doi: 10.1007/s11325-010-0379-7. Epub 2010 Jul 1. PMID 20593281
- [Background] McLaughlin MA, Tamler R, Woodward M, Moline J, Sawit ST, O'Boyle J, Berookhim B, Lu K, Bar-Chama N. Hypogonadism is Independently Associated with Obstructive Sleep Apnea in Middle-aged Men. Poster session presented at: American Heart Association Quality of Care and Outcomes Research 2011 Scientific Sessions; 2011 May 12-14; Washington, DC.
- [Background] Brook RD, Rajagopalan S, Pope CA 3rd, Brook JR, Bhatnagar A, Diez-Roux AV, Holguin F, Hong Y, Luepker RV, Mittleman MA, Peters A, Siscovick D, Smith SC Jr, Whitsel L, Kaufman JD; American Heart Association Council on Epidemiology and Prevention, Council on the Kidney in Cardiovascular Disease, and Council on Nutrition, Physical Activity and Metabolism. Particulate matter air pollution and cardiovascular disease: An update to the scientific statement from the American Heart Association. Circulation. 2010 Jun 1;121(21):2331-78. doi: 10.1161/CIR.0b013e3181dbece1. Epub 2010 May 10. PMID 20458016
- [Background] Clark RN, Green R, Swayze G, et al. Environmental studies of the World Trade Center area after the September 11, 2001 attack. Available at: http://pubs.usgs.gov/of/2001/ofr-01-0429.
- [Background] Landrigan PJ, Lioy PJ, Thurston G, Berkowitz G, Chen LC, Chillrud SN, Gavett SH, Georgopoulos PG, Geyh AS, Levin S, Perera F, Rappaport SM, Small C; NIEHS World Trade Center Working Group. Health and environmental consequences of the world trade center disaster. Environ Health Perspect. 2004 May;112(6):731-9. doi: 10.1289/ehp.6702. PMID 15121517
- [Background] Lioy PJ, Weisel CP, Millette JR, Eisenreich S, Vallero D, Offenberg J, Buckley B, Turpin B, Zhong M, Cohen MD, Prophete C, Yang I, Stiles R, Chee G, Johnson W, Porcja R, Alimokhtari S, Hale RC, Weschler C, Chen LC. Characterization of the dust/smoke aerosol that settled east of the World Trade Center (WTC) in lower Manhattan after the collapse of the WTC 11 September 2001. Environ Health Perspect. 2002 Jul;110(7):703-14. doi: 10.1289/ehp.02110703. PMID 12117648
- [Background] McGee JK, Chen LC, Cohen MD, Chee GR, Prophete CM, Haykal-Coates N, Wasson SJ, Conner TL, Costa DL, Gavett SH. Chemical analysis of World Trade Center fine particulate matter for use in toxicologic assessment. Environ Health Perspect. 2003 Jun;111(7):972-80. doi: 10.1289/ehp.5930. PMID 12782501